CLINICAL TRIAL: NCT00332813
Title: Reducing HIV Risk Among Pregnant Women in Drug Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA020930; R01DA020930 (NIH)
Record Dates: First submitted 2006-06-01; First posted 2006-06-02 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2006-01

CONDITIONS: HIV Risk Behavior
Keywords: HIV Risk Behavior; Pregnancy; Drug Abuse
MeSH Terms: conditions — Substance-Related Disorders

INTERVENTIONS:
Behavioral: HIV Risk Behavior Intervention

SUMMARY:
We propose to develop and pilot test an intervention that addresses both sex- and drug-related HIV risk behavior among pregnant women in drug treatment. In the first phase of the study, we will conduct focus groups with pregnant women in drug treatment, as well as a focus group with their treatment providers, in order to determine key areas of emphasis for an intervention in this population. We will then develop an HIV risk behavior intervention for pregnant women in drug treatment, pilot the intervention with 20 women, and elicit their feedback regarding the intervention. Following refinement of the intervention, we will conduct a small randomized trial (n=60) to examine the impact of the intervention compared to standard care (SC). We expect that, relative to SC, participants randomized to the intervention condition will have lower levels of sex- and drug-related HIV risk behavior.

DETAILED DESCRIPTION:
HIV is a critical and costly health problem for American women. Among pregnant drug abusers, sex- and drug-related HIV risk behavior occur at alarming rates. While motivationally-enhanced HIV risk behavior interventions have demonstrated efficacy with similar populations, very little work has been directed toward pregnant women in drug abuse treatment. The long-term objective of this research program is to reduce HIV risk behavior among pregnant women engaged in drug abuse treatment by developing and establishing the efficacy of an intervention that combines motivational interviewing, psychoeducation, and skill building exercises. Furthermore, we seek to advance knowledge of the mechanism of action by which interventions reduce HIV risk behavior. In the present application, we propose to develop and pilot test an intervention that addresses both sex- and drug-related HIV risk behavior among pregnant women in drug treatment. In the first phase of the study, we will conduct focus groups with pregnant women in drug treatment, as well as a focus group with their treatment providers, in order to determine key areas of emphasis for an intervention in this population. We will then develop an HIV risk behavior intervention for pregnant women in drug treatment, pilot the intervention with 20 women, and elicit their feedback regarding the intervention. Following refinement of the intervention, we will conduct a small randomized trial (n=60) to examine the efficacy of the intervention relative to standard care (SC). We expect that, relative to SC, participants randomized to the intervention condition will have lower levels of sex- and drug-related HIV risk behavior. We will also examine the potential mechanisms by which the intervention produces a reduction in HIV risk behavior. If found to be efficacious, this intervention will help to reduce the acquisition of HIV among pregnant drug abusers, improving health outcomes for the women and their children.Relevance to Public Health: The proposed study is designed to develop and test an intervention to reduce sex- and drug-related behavior that places pregnant drug abusers at risk for HIV infection. If successful, this intervention could reduce the rate of HIV infection in these women and their children.

ELIGIBILITY:
Inclusion Criteria:18 years of age or older, less than 32 weeks gestation, drug dependence (other than nicotine), have engaged in sex- or drug-related HIV risk behaviors at least monthly for 3 months prior to recruitment -

Exclusion Criteria:Currently psychotic, unable to provide names and contact information for two people who could serve as locators

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2006-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Unprotected vaginal or anal intercourse
Sharing of injection drug works

SECONDARY OUTCOMES:
Risk Assessment Battery

CONTACTS AND LOCATIONS:
Overall Officials: Susan E. Ramsey, Ph.D., Principal Investigator — Brown Medical School/Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States